CLINICAL TRIAL: NCT05861843
Title: Craving Assessment in Patients With Alcohol Use Disorder Using Virtual Reality Exposure
Acronym: CRAVE
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Alva Lütt, Dr. med. Alva Lütt, MD, Charite University, Berlin, Germany
Other Study IDs: EA1/190/22
Record Dates: First submitted 2023-04-24; First posted 2023-05-17 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Virtual Reality-based cue exposure paradigm — Virtual Reality (VR) cue exposure to alcohol-associated cues using head-mounted displays (HMD)

SUMMARY:
Alcohol use disorder (AUD) is a burdensome clinical disorder with high relapse rates. Virtual Reality (VR)-based therapeutic and diagnostic approaches have received increasing attention in the treatment of AUD but evidence on the induction of craving via VR scenarios is still needed. Craving for alcohol is associated with psychological and physiological responses. This single-arm clinical study will be conducted including n=60 patients with AUD. Using a head-mounted display (HMD), patients will be confronted with three different VR scenarios (neutral vs. two target situations) while heart rate, heart rate variability (HRV), pupillometry and electrodermal activity (EDA) will be measured continuously. Subjective craving levels will be assessed pre-/during/post-exposure to each VR scenario.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-65 years
* diagnosis of alcohol dependence according to ICD-10 (F10.2)
* completed in-patient withdrawal treatment during the last 3 months
* history of alcohol craving, confirmed via craving questionnaires
* able to provide written informed consent

Exclusion Criteria:

* substance dependence other than alcohol and nicotine
* current alcohol intoxication (randomly tested via measurement of breath alcohol concentration)
* unable to understand the study information, consent form or principles of the study
* abstinence for less than 7 days or on-going consumption of alcohol
* severe neuropsychiatric disorder, e.g. schizophrenia spectrum disorders, bipolar affective disorder or substantial cognitive impairment
* serious illnesses influencing brain-/heart-function with influence on physiological study parameters.
* acute suicidality (or acute endangerment of others)
* concurrent pharmacological treatment targeting AUD (i.e. benzodiazepines) or craving (i.e. acamprosate, disulfiram, naltrexone, nalmefene) and further medication significantly influencing heart frequency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AUD treated in inpatient or outpatient psychiatric clinic
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
change in subjective craving levels elicited by alcohol-associated cues | 20-30 min VR exposure
  Changes in craving levels measured by subjective parameters (visual analogue scale = VAS, scale 0-100) before, during and after VR-exposure to alcohol-associated cues compared to neutral cues
change in psychophysiological craving levels (heart rate) elicited by alcohol-associated cues | 20-30 min VR exposure
  Changes in craving levels measured continuously by heart rate (bpm = beats per minute) during VR-exposure to alcohol-associated cues compared to neutral cues.
change in psychophysiological craving levels (heart rate variability) elicited by alcohol-associated cues | 20-30 min VR exposure
  Changes in craving levels measured continuously by heart rate variability (ms) during VR-exposure to alcohol-associated cues compared to neutral cues.
change in psychophysiological craving levels (electrodermal activity) elicited by alcohol-associated cues | 20-30 min VR exposure
  Changes in craving levels measured continuously by electrodermal activity (micro-Siemens) during VR-exposure to alcohol-associated cues compared to neutral cues.
change in psychophysiological craving levels elicited by alcohol-associated cues | 20-30 min VR exposure
  Changes in craving levels measured continuously by pupillometry (pupil dilation in mm) during VR-exposure to alcohol-associated cues compared to neutral cues.

SECONDARY OUTCOMES:
context-related change in craving levels | 20-30 minutes VR Exposure
  changes in subjective and objective craving levels compared between the two VR-scenarios bar vs. living room
development of subjective craving levels post-exposure | 3 hours after VR-exposure
  changes of subjective craving (VAS) over the following 3 hours after VR-exposure

CONTACTS AND LOCATIONS:
Overall Officials: Alva Lütt, Dr. med., Principal Investigator — Psychiatrische Universitätsklinik der Charité im St. Hedwig Krankenhaus, 10115 Berlin, Germany
Locations (1):
- Psychiatric University Hospital Charité at St. Hedwig Hospital, Berlin, Germany

REFERENCES:
- [Derived] Lutt A, Tsamitros N, Wolbers T, Rosenthal A, Brocker AL, Schoneck R, Bermpohl F, Heinz A, Beck A, Gutwinski S. An explorative single-arm clinical study to assess craving in patients with alcohol use disorder using Virtual Reality exposure (CRAVE)-study protocol. BMC Psychiatry. 2023 Nov 14;23(1):839. doi: 10.1186/s12888-023-05346-y. PMID 37964300